CLINICAL TRIAL: NCT03898934
Title: Dose Vitamin-D Supplementation Affect Reproductive Outcomes in Patients With Polycystic Ovary Syndrome?
Brief Title: Vitamin D Supplementation in PCOS Patients
Acronym: PCOvit-D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCOvit-D
Record Dates: First submitted 2019-03-30; First posted 2019-04-02 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: PCOS
Keywords: PCOS; Vitamin D; Supplementation; Ovulation; Pregnancy
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: The 2 groups will be treated at the same time
Who Masked: Participant, Care Provider
Masking Description: Both patients and gynecologists were binded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental): These patients will receive 6000IU daily for 8 weeks then 2000IU maintenance till pregnancy or end of study
  Interventions: Drug: Vitamin D
- Placebo group (Placebo Comparator): These group will receive placebo for the same periods of study group
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Vitamin D — receive 6000iu daily for 8 weeks
  Arms: Vitamin D group
Drug: Placebo Oral Tablet — placebo for the same period
  Arms: Placebo group

SUMMARY:
To assess whether Vitamin D supplementations for patients with polycystic ovary syndrome in conjunction with clomiphene citrate are beneficial or not

DETAILED DESCRIPTION:
This study is double blinded randomized controlled study conducted at Tanta University hospitals in the period from April 2019 to March 2022. Patients and methods: One hundred twelve patients were recruited and randomly allocated into 2 groups; study group with Vitamin D supplementation and control group without Vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

* PCOS
* Infertile
* Vitamin D deficient

Exclusion Criteria:

* Age less than 20 and more than 35
* Non PCOS patients
* Obese patients
* Previous ovarian surgery
* Previous oophrectomy of one ovary

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Ovulation rate | 3 months
  Number of mature follicles obtained
Pregnancy rate | 3 months
  Number of patients who get pregnant

CONTACTS AND LOCATIONS:
Locations (1):
- Ayman Shehata Dawood, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share results
Supporting Information: Study Protocol
Time Frame: 3 months